CLINICAL TRIAL: NCT03021746
Title: Fostering Sustainability Through Diabetes Self-Management Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gretchen Piatt, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00104965
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus
Keywords: African-American
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Parish Nurse plus Peer Leader (Experimental): The focus of this approach is for Peer Leaders (PL) to provide Diabetes Self Management Support (DSMS) with the oversight of Parish Nurses (PN). The first component starts with group-based Diabetes Self Management Education (DSME) provided by Certified Diabetes Educators (CDE), co-facilitated by PN and PL and held at the church. PL will also facilitate activities including behavioral goal setting, monthly phone contacts, and preparation for a diabetes-related health care visit, with oversight of PN. As the study progresses, PL and PN will have progressive leadership responsibilities. Following DSME, participants will be invited to attend 12 months of monthly DSMS support groups led by the PL, with oversight from the PN. This approach allows for PN to provide direct supervision to PL in areas of clinical content, educational methods, and group facilitation and communication skills.
  Interventions: Behavioral: Diabetes Self Management Support (DSMS)
- Peer Leader Only (Experimental): This approach will contain the same elements as the PN plus PL approach, except that a PN will not be used. Rather, PL will provide all aspects of DSMS, including behavioral goal setting, monthly phone contacts, and preparation for a diabetes-related health care visit. This approach will be delivered in a group setting. DSME will be provided by CDEs and co-facilitated by a PL to ensure consistency in the DSME content. Following DSME, participants will be invited to attend 12 monthly DSMS groups led by PL. Following the group sessions, participants will transition into a period of ongoing support. During this time, participants and PL will be encouraged to foster DSMS through programs and initiatives that are meaningful to them, utilizing the existing church infrastructure. If needed, PL may contact the CDE for additional information
  Interventions: Behavioral: Diabetes Self Management Support (DSMS)
- Parish Nurse Only (Experimental): The main focus of this approach will contain all of the same elements as the PN plus PL approach, except that PL will not be used. Rather, the PN will provide all aspects of Diabetes Self Management Support (DSMS), including facilitation of goal setting, monthly phone contacts, and preparation for a diabetes-related health care visit. Diabetes Self Management Education (DSME) will be provided by CDEs and co-facilitated by a PN to ensure consistency in the DSME content. Following DSME, participants will be invited to attend 12 months of monthly, DSMS support groups led by the PN. Following support sessions, participants will transition into a period of ongoing support, where the participants and PN will be encouraged to continue to foster DSMS through programs and initiatives that are meaningful to them, utilizing the existing church infrastructure. The PN may answer clinical questions and may contact the CDE for additional information if needed.
  Interventions: Behavioral: Diabetes Self Management Support (DSMS)

INTERVENTIONS:
Behavioral: Diabetes Self Management Support (DSMS)

SUMMARY:
To understand the effectiveness of three approaches to address diabetes self-management support compared to enhanced usual care in church-based settings.

DETAILED DESCRIPTION:
To understand the effectiveness of three approaches to address diabetes self-management support compared to enhanced usual care in church-based settings.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 diabetes for at least 6 months
* Be Black/African American
* Be a resident of metro-Detroit, Toledo, or Flint
* Be at least 21 years old
* Be under the care of a physician for diabetes
* Have transportation to attend the program

Exclusion Criteria:

* Have Type 2 diabetes for less than 6 months
* Under 21 years of age
* Not under care of physician
* Lack of transportation to attend the program

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2016-03; Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in A1C Blood Glucose level | During this study, A1c will be measured at five time points; baseline, 6 months, 9 months, 21 months, and 33 months.
  An A1C test is a blood test that reflects one's average blood glucose levels over the previous 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Piatt, MPH, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No